CLINICAL TRIAL: NCT04820049
Title: F573 for Injection Phase Ia Clinical Trial.
Brief Title: F573 Ia Clinical Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Continent Pharmaceutical Co, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GNI-F573-202001
Record Dates: First submitted 2021-02-03; First posted 2021-03-29 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2021-03

CONDITIONS: Tolerance; Pharmacokinetic
MeSH Terms: interventions — benzyloxycarbonyl-valyl-aspartic acid fluoromethyl ketone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator)
  Interventions: Other: Placebo
- F573 group (Experimental)
  Interventions: Drug: F573

INTERVENTIONS:
Drug: F573 — F573 for injection
  Arms: F573 group
Other: Placebo — Water for injection
  Arms: Placebo group

SUMMARY:
Tolerance and PK study of F573

DETAILED DESCRIPTION:
The tolerance and PK study of single dose and multi dose F573.

ELIGIBILITY:
Inclusion criteria (each item must be met)

1. Healthy volunteers, male and female;
2. Age: 18-45 years old;
3. Weight: male ≥50kg, female ≥45kg, 19≤BMI≤26 (BMI= weight (kg)/height 2 (m2));
4. Passed the comprehensive physical examination, that is, the routine blood and urine, blood pregnancy, blood glucose, blood lipids, blood electrolytes, hepatitis B surface antigen, liver and kidney function, hepatitis C, HIV and syphilis antibody test, electrocardiogram, cigarette test, urine drug screening, alcohol breath test, chest X-ray and other abnormal or abnormal without clinical significance;
5. Have a detailed understanding of the nature, significance, possible benefits, possible inconveniences and potential risks of the trial before the study, and voluntarily participate in the clinical trial, be able to communicate well with the researchers, comply with the requirements of the whole study, and have the ability to understand and sign the written informed consent.

Exclusion criteria (if one of them is met)

1. Participated in any other clinical trials within the three months prior to the trial;
2. (preliminary) of any process may affect test security, or drug in the body of the disease, including but not limited to: heart, liver, kidney, endocrine, the digestive tract, immune system and respiratory system always or the existing system diseases (especially cardiovascular diseases including cardiovascular disease risk, any impact on drug absorption of gastrointestinal diseases (such as irritable bowel syndrome, inflammatory bowel disease), active pathological bleeding (such as peptic ulcer), urticaria, eczema, dermatitis, epilepsy, allergic rhinitis, asthma, etc.);
3. (Inquiry) Allergic constitution: if there is a history of drug, food allergy or skin allergy;
4. (Inquiry) Use of any drug that inhibits or induces liver metabolism to the drug within 28 days prior to use of the study drug (Common liver enzyme inducers: barbiturates such as phenobarbital, carbamazepine, aminomide, griseofulvin, metalpropanol, phenytoin, glumide, rifampicin, dexamethasone; Common liver enzyme inhibitors: chlorpromazine, cimetidine, ciprofloxacin, metronidazole, chloramphenicol, isoniazid, sulfonamides);
5. Have used any medicine (including Chinese herbal medicine) and health care products within 14 days before the first administration;
6. (Consultation) People who have special requirements for food and cannot abide by the unified diet (such as intolerance to standard food);
7. (consultation) can not tolerate venipuncture, intramuscular injection and/or have a history of dizziness of blood and needles;
8. (Consultation) Drinking excessively tea, coffee or caffeinated beverages for a long time in the past (more than 8 cups a day, 1 cup =250mL); Or study within 48 hours before the first administration of the drug, the intake of any food or beverage containing caffeine (such as coffee, strong tea, chocolate, etc.) and other special diet that affects the absorption, distribution, metabolism, excretion of the drug;
9. (Inquiry) Previous alcohol abuse (i.e., more than 28 SUs per week for men and more than 21 SUs per week for women (1 SU contains 14 g of alcohol, such as 360 mL beer or 45 mL 40% spirits or 150 mL wine); Or regular alcohol consumption (more than 14 standard units per week) in the 6 months prior to the study; Or have taken any alcoholic product within 24 hours prior to first administration;
10. (Inquiry) who donated blood or suffered massive bleeding (greater than 450 mL) within 3 months before the first administration of the study, or who planned to donate blood or blood components during the study or within 3 months after the end of the study;
11. (Inquiry) Acute disease occurs in the pre-study screening stage or before the study medication;
12. (Inquiry) Those who took food or beverage (such as grapefruit, mango, dragon fruit, grape juice, orange juice and other rich flavonoids or citrus compounds) containing enzymes that can induce or inhibit liver metabolism within 24 hours before the first administration of medication;
13. (Consultation) had surgery within 3 months prior to the screening period, or planned to have surgery during the study period;
14. (Inquiry) Previous history of drug abuse; With a history of drug abuse;
15. Smoking more than 5 cigarettes per day in the 14 days before screening, or unable to stop using any tobacco products during the trial;
16. Screening (Consultation) Those who smoked or used any tobacco products during the admission period;
17. Positive results of nicotine test;
18. Alcohol breath test with test results greater than 0.0mg/100mL;
19. Positive urine drug screening;
20. Pregnant or lactating women;
21. Those who had family planning during the study period and within 6 months after the end of the study;
22. Refusing to use non-drug contraception during the study period
23. novel coronavirus nucleic acid test positive or antibody test positive;
24. The investigator considers that there is any circumstance that may affect the subject's ability to give informed consent or follow the study protocol, or that the participant's participation in the study may affect the study result or their own safety.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-11-06 (Actual)

PRIMARY OUTCOMES:
MTD of F573 in health people | up to 7 days
Cmax of F573 in health people | up to 7 days
Tmax of F573 in health people | up to 7 days
t1/2 of F573 in health people | up to 7 days
AUC of F573 in health people | up to 7 days

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 8 days

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No